CLINICAL TRIAL: NCT06647576
Title: Abbott Neurosphere™ Pilot Study: Remote Monitoring and Virtual Clinic Features in Improving Quality of Life and Potential Cost-Saving
Brief Title: Exploring Neurosphere's Remote Monitoring and Virtual Clinic Features in Improve Quality of Life and Reduce Costs
Acronym: TRC-AB-1
Status: Enrolling by invitation | Type: Observational
Sponsor: Mahesh Pattabiraman (Industry)
Responsible Party: Sponsor-Investigator, Mahesh Pattabiraman, Chief Executive, TriCity Research Center
Organization: TriCity Research Center (Industry)
Other Study IDs: IIS-24-ABT-001
Record Dates: First submitted 2024-10-14; First posted 2024-10-18 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Chronic Neuropathic Pain; Chronic Pain Management; Spinal Cord Stimulation (SCS); Pain Modulation; Failed Back Surgery Syndrome
Keywords: chronic pain; spinal cord stimulation; neuropathic pain; Remote Pain Management; BurstDR Technology; Chronic Pain in Rural Populations
MeSH Terms: conditions — Failed Back Surgery Syndrome; Chronic Pain; Neuralgia | interventions — Spinal Cord Stimulation; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Test: Patients receiving SCS therapy through Neutrosphere virtual clinic platform (remote pain management group).
  Interventions: Device: Spinal Cord Stimulation - Neurosphere
- Control Group: Participants in this group will receive traditional in-person care for their SCS therapy. Group regular clinic visits for therapy adjustments, monitoring, and pain management
  Interventions: Device: Spinal Cord Stimulation - In Clinic

INTERVENTIONS:
Device: Spinal Cord Stimulation - In Clinic — Control Group Intervention: In-Person SCS therapy. Device settings, such as pulse width and frequency, will be adjusted during regular clinic visits. Follow-up assessments for pain relief, quality of life, and therapy effectiveness will occur at 1, 3, and 6-month intervals over a 6-month period.
  Other Names: neuromodulation; In Person SCS
  Groups: Control Group
Device: Spinal Cord Stimulation - Neurosphere — Test Group Intervention: Test group participants will receive remote monitoring and therapy adjustments through the Neurosphere™ virtual clinic platform. Participants in test group will have trial and end of trial phases in clinic, but further SCS therapy will be performed through Neurosphere. Clinicians will adjust the SCS device settings, including pulse width and burst frequency, remotely. This intervention allows patients to avoid in-person visits while receiving continuous, personalized care, with follow-up assessments at 1, 3, and 6 months over a 6-month period.
  Other Names: Remote Pain Management
  Groups: Test

SUMMARY:
This study evaluates the effectiveness of Abbott's Proclaim™ and Eterna™ Spinal Cord Stimulator (SCS) systems, along with the Neurosphere™ virtual clinic platform, in managing chronic pain. The goal is to assess how remote monitoring and virtual care can improve pain relief and reduce healthcare costs compared to traditional in-person care. Adults with chronic pain will either receive treatment through in-person visits or remotely using Neurosphere™. The study will measure pain relief, quality of life, and healthcare expenses over six months, aiming to improve access to pain management, especially for patients in rural areas.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years and older experiencing chronic neuropathic pain that is refractory to medical treatment and eligible for SCS based on FDA-approved indications.
* Individuals who can legally provide informed consent.

Exclusion Criteria:

* Patients unable or unwilling to adhere to the requirements of remote monitoring, follow-up schedules, or other aspects of the study protocol.
* Patients with uncontrolled psychiatric conditions, including severe depression or anxiety, which could interfere with their ability to participate fully in the study or accurately report outcomes.
* Women who are currently pregnant or breastfeeding, as the safety and efficacy of SCS in these populations are not established.
* Patients who have previously experienced significant adverse events or complications from SCS implantation or stimulation that would make further use unsafe or ineffective.
* Patients with other active implantable devices (e.g., pacemakers or defibrillators) that could interfere with the functionality of the SCS system.
* Patients with a documented history of substance abuse within
* Patients with significant comorbid conditions (severe cardiovascular disease, unmanaged diabetes, uncontrolled infection, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult participants aged 19 years and older who are experiencing chronic neuropathic pain that is refractory to medical treatment and are eligible for SCS therapy based on FDA-approved indications. Participants will be recruited from a rural population, with effort made for including individuals from diverse socioeconomic backgrounds. Study will enroll patients who can legally provide consent and are willing to adhere to the study protocol, including remote monitoring or in-person follow-up visits.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Pain Relief - NRS | Baseline, 1 month, 3 months, and 6 months post-intervention
  Pain relief in numerical pain rating scale (NRS). Numerical points.
Quality of Life and Functional Disability Improvements - ODI | Baseline, 1 month, 3 months, and 6 months post-intervention
  Change in quality of life and functional disability in participants quantified through numerical response to Oswestry Disability Index (ODI) compared to baseline
Healthcare Cost Reduction | From baseline to 6 months post-intervention
  This outcome measures the reduction in healthcare costs associated with the use of the Neurosphere™ remote monitoring platform compared to traditional in-person care. Costs will be assessed through an analysis of healthcare resource utilization using time-driven activity-based costing TDABC methodology.

CONTACTS AND LOCATIONS:
Locations (1):
- Grand Island Pain Relief Center, Grand Island, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD related to the primary and secondary outcomes of the study, including anonymized data on pain relief, quality of life, healthcare utilization, and cost-effectiveness, will be shared. The shared data will include patient-reported outcomes (e.g., ODI and NRS for pain), as well as relevant clinical and financial data collected throughout the study. A detailed data dictionary, explaining all variables, will be provided to ensure proper interpretation. IPD will be made available upon reasonable request after publication of the study results
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code